CLINICAL TRIAL: NCT02908477
Title: DART-HPV: A Phase III Evaluation of De-escalated Adjuvant Radiation Therapy for HPV-Associated Oropharynx Cancer
Brief Title: Evaluation of De-escalated Adjuvant Radiation Therapy for Human Papillomavirus (HPV)-Associated Oropharynx Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-004083; MC1675 (Other: Mayo Clinic in Rochester); NCT03421470 (obsolete NCT alias)
Record Dates: First submitted 2016-08-26; First posted 2016-09-21 (Estimated); Results first posted 2024-04-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Oropharynx Cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- De-escalated Adjuvant Radiation Therapy (Experimental): Docetaxel 15 mg/m2 days 1, 8 + Radiation Therapy (RT) 30 Gy/1.5 Gy fractions twice daily (b.i.d.) days 1-12 only (intermediate risk) or 36 Gy/1.8 Gy b.i.d. fractions (high risk)
  Interventions: Radiation: Adjuvant Radiation Therapy; Drug: Docetaxel
- Standard of Care Treatment (Active Comparator): RT 60 Gy/2 Gy fractions daily (qday) days 1-40. For high risk, add weekly Cisplatin 40 mg/m2 (Around days 1, 8, 15, 22, 29, 36)
  Interventions: Radiation: Adjuvant Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: Adjuvant Radiation Therapy — 60 Gy / 2 Gy fractions (standard arm) 30 - 36 Gy / 1.5 - 1.8 Gy b.i.d. fractions (experimental arm)
Drug: Docetaxel — 15 mg/m2. Experimental arm only.
  Other Names: Taxotere
  Arms: De-escalated Adjuvant Radiation Therapy
Drug: Cisplatin — 40 mg/m2. Standard arm only.
  Other Names: cisplatinum
  Arms: Standard of Care Treatment

SUMMARY:
This study is designed for patients with a cancer of the oropharynx (tonsils or base of tongue) caused by the HPV virus. Traditional treatment involves surgery followed by six weeks of daily radiation therapy. This study investigates a less intense radiation treatment following surgery that uses half the dose of radiation given over two weeks rather than six weeks. Patients will be randomly assigned to receive the less intense treatment versus the traditional treatment by coin flip. Patients are twice as likely to receive the less intense treatment during randomization.

DETAILED DESCRIPTION:
Recent studies suggest that tumors in the oropharynx (tonsils or base of tongue) caused by the HPV virus are much more sensitive to radiation and chemotherapy. Standard treatment for HPV associated oropharynx tumor after surgery involves six weeks of radiation therapy and has many long term side effects and complications.

Mayo Clinic recently piloted a study investigating whether patients with HPV-associated oropharynx tumors can receive less radiation and chemotherapy after surgery when compared with the standard treatment. The investigators current study will compare the new, shorter treatment course (2 weeks of treatment) with the standard course of treatment (six weeks). Patients will be randomized to either the less intense or standard treatment arm. Patients will be twice as likely to receive the less intense treatment during randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histological confirmation of HPV+ squamous cell carcinoma of the oropharynx. HPV positivity will be defined as positive staining for p16 on immunohistochemistry (IHC).
* Gross total surgical resection with curative intent of the primary tumor and at least unilateral neck dissection within 7 weeks of registration.
* ECOG Performance Status (PS) 0 or 1
* Absence of distant metastases on standard diagnostic work-up ≤ 10 weeks prior to registration. (Chest CT, Chest x-ray (CXR), or PET/CT.)
* Must have one of the following risk factors:

  * Lymph node > 3 cm
  * 2 or more positive lymph nodes
  * Perineural invasion
  * Lymphovascular space invasion
  * T3 or T4 primary disease
  * Lymph node extracapsular extension
* The following laboratory values obtained ≥14 days prior to registration.

  * Absolute neutrophil count (ANC) ≥1500/mm3
  * Platelet count ≥100,000/mm3
  * Hemoglobin ≥8.0g/dL
  * Creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min
  * Total bilirubin < 2 x institutional upper limit of normal (ULN)
  * AST or ALT < 3 x institutional ULN
* Negative pregnancy test done ≤7 days prior to registration, for women of childbearing potential only.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Provide informed written consent.
* Willingness to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study).

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
* Immunocompromised patients and patients known to be HIV positive.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm.
* Other active malignancy ≤ 5 years prior to registration. EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix. NOTE: If there is a history or prior malignancy, they must not be receiving other specific treatment for their cancer.
* Prior history of radiation therapy to the affected site.
* History of connective tissue disorders such as rheumatoid arthritis, lupus, or Sjogren's disease.
* Presence of any of the following risk factors after surgery:

  * Any positive surgical margin.
  * Adenopathy below the clavicles
* Prior systemic chemotherapy.
* Receiving any medications or substances which in the opinion of the investigators would interfere with treatment. Examples could include strong inhibitors of CYP3A4 at oncologist discretion (see Appendix IV).
* Severe pre-existing ototoxicity or neuropathy that would, in the opinion of the investigator, preclude the use of cisplatin chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2024-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ma, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma D, Price K, Moore E, Patel S, Hinni M, Routman D, Fruth B, Foster N, Van Abel K, Yin L, Neben-Wittich M, Garces Y, McGee L, Lester S, Rwigema JC, Holtzman A, Price D, Janus J, Kasperbauer J, Chintakuntlawar A, Garcia J, Foote R. De-escalated adjuvant radiotherapy versus standard adjuvant treatment for human papillomavirus-associated oropharyngeal squamous cell carcinoma (MC1675): a phase 3, open-label, randomised controlled trial. Lancet Oncol. 2025 Sep;26(9):1227-1239. doi: 10.1016/S1470-2045(25)00324-9. PMID 40907518
- [Derived] Routman DM, Van Abel KM, Price KA, Moore EJ, Patel SH, Hinni ML, Fruth B, Foster NR, Yin LX, Neben-Wittich M, Garces YI, McGee LA, Lester SC, Gamez ME, Rwigema JM, Holtzman AL, Price DL, Janus JR, Kasperbauer JL, Chintakuntlawar AV, Garcia JJ, Foote RL, Ma DJ. ctDNA and Recurrence Risk for Adjuvant De-Escalation in HPV-Positive Oropharyngeal Carcinoma: A Secondary Analysis of the DART Phase 3 Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2025 Jul 1;151(7):665-672. doi: 10.1001/jamaoto.2025.0903. PMID 40402484

RESULTS

PARTICIPANT FLOW:
Groups:
- De-escalated Adjuvant Radiation Therapy (DART): Docetaxel 15 mg/m2 days 1, 8 and Radiation Therapy (RT) 30 Gy/1.5 Gy fractions twice daily (b.i.d.) days 1-12 only (intermediate risk) or 36 Gy/1.8 Gy b.i.d. fractions (high risk)> > Adjuvant Radiation Therapy: 60 Gy / 2 Gy fractions (standard arm)> 30 - 36 Gy / 1.5 - 1.8 Gy b.i.d. fractions (experimental arm)>
  > Docetaxel: 15 mg/m2. Experimental arm only.
- Standard of Care Treatment (SOC): RT 60 Gy/2 Gy fractions daily (qday) days 1-40. > For high risk, add weekly Cisplatin 40 mg/m2 (Around days 1, 8, 15, 22, 29, 36)> > Adjuvant Radiation Therapy: 60 Gy / 2 Gy fractions (standard arm)> 30 - 36 Gy / 1.5 - 1.8 Gy b.i.d. fractions (experimental arm)>
  > Cisplatin: 40 mg/m2. Standard arm only.
Period: Overall Study
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC)
Started | 136 | 92
Completed | 128 | 64
Not Completed | 8 | 28
Not completed — Withdrawal by Subject | 8 | 28

BASELINE CHARACTERISTICS:
Population: All registered patients
Groups:
- Total: Total of all reporting groups
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC) | Total
Number analyzed (Participants) | 136 | 92 | 228
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 81] | 58 [35 to 73] | 59 [35 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 121 | 81 | 202
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 123 | 84 | 207
  Unknown or Not Reported | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 128 | 87 | 215
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Grade 3+ Adverse Events Rate
Description: To compare rate of late grade 3-5 toxicities between de-escalated adjuvant radiation therapy (DART) and standard adjuvant therapy.
Time Frame: 2 years
Population: All treated patients
Measure: Number; unit: events per participant
Groups:
- De-escalated Adjuvant Radiation Therapy (DART): Docetaxel 15 mg/m2 days 1, 8 and Radiation Therapy (RT) 30 Gy/1.5 Gy fractions twice daily (b.i.d.) days 1-12 only (intermediate risk) or 36 Gy/1.8 Gy b.i.d. fractions (high risk)
  >
  > Adjuvant Radiation Therapy: 60 Gy / 2 Gy fractions (standard arm)
  > 30 - 36 Gy / 1.5 - 1.8 Gy b.i.d. fractions (experimental arm)
  >
  > Docetaxel: 15 mg/m2. Experimental arm only.
- Standard of Care Treatment (SOC): RT 60 Gy/2 Gy fractions daily (qday) days 1-40. > For high risk, add weekly Cisplatin 40 mg/m2 (Around days 1, 8, 15, 22, 29, 36)
  >
  > Adjuvant Radiation Therapy: 60 Gy / 2 Gy fractions (standard arm)
  > 30 - 36 Gy / 1.5 - 1.8 Gy b.i.d. fractions (experimental arm)
  >
  > Cisplatin: 40 mg/m2. Standard arm only.
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC)
Number analyzed (Participants) | 130 | 64
events per participant | .032 | .115

2. Secondary Outcome: Local/Regional Control
Description: Local/regional failure percentage as assessed by imaging or physical exam at 2 years after study registration for patients treated with DART vs standard therapy.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC)
Number analyzed (Participants) | 130 | 64
percentage of participants | 95.9 | 98.3

3. Secondary Outcome: Quality of Life Between DART and Standard Adjuvant Therapy - FACT-HN
Description: To compare the overall QOL between DART and standard adjuvant therapy at 1-year post-treatment as measured by the Functional Assessment of Cancer Therapy - Head & Neck (FACT-HN) questionnaire. The FACT-HN consists of 12 questions related to symptoms and feeling over the past 7 days. Items are answered on a scale of 0-4 where 0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, and 4=very much.
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Quality of Life Between DART and Standard Adjuvant Therapy - EORTC-QLQ-HN35
Description: To compare the overall QOL between DART and standard adjuvant therapy at 1-year post-treatment as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Head and Neck Module (EORTC-QLQ-HN35). The questionnaire consists of 35 items related to symptoms or problems during the past week. Thirty (30) items are answered on a scale of 0-4 where 0=not at all; 1=a little; 3=quite a bit, and 4=very much, and five (5) items are answered with yes/no.
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Overall Survival
Description: Percentage of patients alive at 2 years.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC)
Number analyzed (Participants) | 130 | 64
percentage of participants | 96.9 | 98.3

6. Secondary Outcome: Disease-free Survival
Description: Percentage of patients disease free and alive at 2 years.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC)
Number analyzed (Participants) | 130 | 64
percentage of participants | 88.2 | 96.6

7. Secondary Outcome: Distant Failure Associated With DART vs Standard Treatment
Description: Distant failure is defined as cancer that has recurred or spread to a part of the body far away from the original tumor site
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected over 2 years and mortality was collected over 5 years
Groups:
- De-escalated Adjuvant Radiation Therapy (DART): Docetaxel: 15 mg/m2. Experimental arm only.
- Standard of Care Treatment (SOC): Cisplatin: 40 mg/m2. Standard arm only.
Arm/Group | De-escalated Adjuvant Radiation Therapy (DART) | Standard of Care Treatment (SOC)
All-Cause Mortality (participants affected / at risk) | 2/136 | 9/92
Serious Adverse Events (participants affected / at risk) | 0/136 | 1/92
Other Adverse Events (participants affected / at risk) | 128/136 | 60/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | De-escalated Adjuvant Radiation Therapy (DART) (N=136) | Standard of Care Treatment (SOC) (N=92)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | De-escalated Adjuvant Radiation Therapy (DART) (N=136) | Standard of Care Treatment (SOC) (N=92)
Accessory nerve disorder (Nervous system disorders) | 27 (27) | 13 (13)
Alopecia (Skin and subcutaneous tissue disorders) | 25 (25) | 17 (17)
Anxiety (Psychiatric disorders) | 31 (31) | 20 (20)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (6)
Brachial plexopathy (Nervous system disorders) | 10 (10) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 48 (48) | 36 (36)
Depression (Psychiatric disorders) | 19 (19) | 16 (16)
Dermatitis radiation (Injury, poisoning and procedural complications) | 98 (98) | 57 (57)
Dry mouth (Gastrointestinal disorders) | 128 (128) | 60 (60)
Dysarthria (Nervous system disorders) | 12 (12) | 8 (8)
Dysesthesia (Nervous system disorders) | 56 (56) | 25 (25)
Dysgeusia (Nervous system disorders) | 124 (124) | 57 (57)
Dysphagia (Gastrointestinal disorders) | 116 (116) | 58 (58)
Ear pain (Ear and labyrinth disorders) | 20 (20) | 15 (15)
Edema face (General disorders) | 18 (18) | 12 (12)
Esophagitis (Gastrointestinal disorders) | 49 (49) | 25 (25)
Facial nerve disorder (Nervous system disorders) | 7 (7) | 1 (1)
Fatigue (General disorders) | 124 (124) | 60 (60)
Fibrosis deep connect tissue (Musculoskeletal and connective tissue disorders) | 98 (98) | 51 (51)
Hearing impaired (Ear and labyrinth disorders) | 19 (19) | 16 (16)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 45 (45) | 29 (29)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Lymphedema (Vascular disorders) | 73 (73) | 46 (46)
Malaise (General disorders) | 13 (13) | 7 (7)
Mucosal infection (Infections and infestations) | 30 (30) | 13 (13)
Mucositis oral (Gastrointestinal disorders) | 98 (98) | 51 (51)
Nausea (Gastrointestinal disorders) | 34 (34) | 29 (29)
Neck edema (General disorders) | 66 (66) | 50 (50)
Oral pain (Gastrointestinal disorders) | 97 (97) | 49 (49)
Pain (General disorders) | 101 (101) | 54 (54)
Pain of skin (Skin and subcutaneous tissue disorders) | 9 (9) | 29 (29)
Paresthesia (Nervous system disorders) | 73 (73) | 38 (38)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 31 (31) | 21 (21)
Salivary duct inflammation (Gastrointestinal disorders) | 93 (93) | 47 (47)
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 101 (101) | 50 (50)
Trismus (Musculoskeletal and connective tissue disorders) | 33 (33) | 28 (28)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 53 (53) | 31 (31)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6)
Weight loss (Investigations) | 47 (47) | 40 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT02908477/Prot_SAP_000.pdf